CLINICAL TRIAL: NCT06576830
Title: Single-Dose Intraoperative Methadone for Pain Management in Pediatric Tonsillectomy: A Randomized Double Blind Clinical Trial
Brief Title: Optimization of Pediatric Tonsillectomy to IMprove AnaLgesia
Acronym: OPTIMAL
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00114677; 1R01HD114678-01 (NIH)
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Pain, Postoperative; Tonsillar Hypertrophy; Tonsillitis; Pediatric Sleep Apnea; Sleep-Disordered Breathing
Keywords: Methadone; Tonsillectomy; Opioid
MeSH Terms: conditions — Pain, Postoperative; Tonsillitis; Sleep Apnea Syndromes | interventions — Methadone; Fentanyl; Hydromorphone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Short acting opioids: Fentanyl/Hydromorphone (Active Comparator): Per Routine Care
  Interventions: Drug: Fentanyl/Hydromorphone
- Long acting opioid: Methadone (Active Comparator): Initial Dosing: 0.15 mg/kg age-ideal body weight in children age 3 - < 12 years and 0.2 mg/kg age-ideal body weight in adolescents age 12 - 17 years.
  Dose escalation (possible, based on interim analysis): 0.2 mg/kg age-ideal body weight in children age 3 - < 12 years and 0.25 mg/kg age-ideal body weight in adolescents age 12 - 17 years.
  Interventions: Drug: Methadone

INTERVENTIONS:
Drug: Methadone — Single-dose intraoperative intravenous methadone with initial dose at 0.15 mg/kg in children and 0.2 mg/kg in adolescents.
  Arms: Long acting opioid: Methadone
Drug: Fentanyl/Hydromorphone — Per routine care, given as needed
  Arms: Short acting opioids: Fentanyl/Hydromorphone

SUMMARY:
The purpose of this study is to compare the use of short acting opioids (fentanyl/hydromorphone) with long acting opioids (methadone) for pain control following tonsillectomy surgery in children and adolescents.

DETAILED DESCRIPTION:
This is a randomized, double-blind, parallel-group, dose-escalation investigation. Participants ("children" defined as ages 3 - < 12 years and "adolescents" defined as ages 12 - 17 years) will be randomized 2:1 to either methadone or short-acting opioid. Surgical and anesthesia care, except for intraoperative opioid management, are not altered for study purposes. The trial will include 2 periods in 3 parallel age groups. In the first period, each age cohort will recruit 66 patients (44 methadone, 22 control). Children will be randomized to methadone 0.15 mg/kg age-ideal body weight and adolescents to 0.2 mg/kg age-ideal body weight. When an age cohort reaches 66 patients, this is the end of the first period. At that time, an unblinded interim analysis will be conducted in that cohort to determine if dose escalation to 0.2 mg/kg dose in children and the 0.25 mg/kg dose in adolescents are met. Methadone dose escalation will be based on clinically meaningful differences in need for rescue opioid in the PACU and the absence of well-defined opioid adverse events. Outcomes data will be collected in hospital and after discharge. With daily surveys for 7 days, and 3 phone calls on day 30, 3 months and 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 3 and < 18 years
2. Elective tonsillectomy +/- adenoidectomy
3. Signed informed consent by parent or legal guardian
4. Children >= 12 years must provide signed written consent, Children >= 7 years must provide verbal assent
5. Negative pregnancy test within 48 hours for post pubescent females

Exclusion Criteria:

1. History of chronic kidney or liver disease
2. Current diagnosis of a chronic pain disorder
3. Planned admission to the Pediatric Intensive Care Unit (PICU)
4. Additional procedures under general anesthesia for which opioids would be prescribed

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 440 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who required rescue opioid administration in the PACU (post-anesthesia care unit) | Up to 6 hours post surgery
  Binary (yes/no) need for opioid in the PACU

SECONDARY OUTCOMES:
Total amount of opioid medication administered | Up to 7 days post surgery
  Postoperative opioid use expressed in morphine milligram equivalents per kilogram
Opioid administration in the PACU (post-anesthesia care unit) | Up to 6 hours post surgery
  Postoperative opioid use in the recovery room expressed in morphine milligram equivalents per kilogram
Opioid administration post PACU (post-anesthesia care unit) | Up to 7 days post surgery
  Postoperative opioid use after PACU discharge expressed in morphine milligram equivalents per kilogram
Evaluation of participant's pain as measured by Numeric Pain Rating Scale | Up to 7 days post surgery
  Numeric Pain Rating Scale, 0-10. 0 no pain, 10 worst possible pain
Number of participants with adverse event in the PACU (post-anesthesia care unit) | Up to 6 hours post surgery
  Adverse events will only include those that are determined to be related to the study drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M. Einhorn, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared in the NICHD DASH repository.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Per NIH guidelines. Data will be available indefinitely.
Access Criteria: NICHD DASH
URL: https://dash.nichd.nih.gov/

REFERENCES:
- [Background] Einhorn LM, Hoang J, La JO, Kharasch ED. Single-dose Intraoperative Methadone for Pain Management in Pediatric Tonsillectomy: A Randomized Double-blind Clinical Trial. Anesthesiology. 2024 Sep 1;141(3):463-474. doi: 10.1097/ALN.0000000000005031. PMID 38669011